CLINICAL TRIAL: NCT04177173
Title: Comparison of Combination of Methotrexate and Statins With Methotrexate Alone as an Anti-inflammatory Agent in the Treatment of Rheumatoid Arthritis.
Brief Title: Methotrexate and Statins With Methotrexate Alone in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Rabia Rathore, Associate Professor of Medicine, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5181/REG./KEMU/2017
Record Dates: First submitted 2019-04-07; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Methotrexate; Statins; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Simvastatin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin & Methotrexate (Experimental): Methotrexate 10 mg once a week per oral for 6 months and Statins (Simvastatin) 20 mg once a day per oral
  Interventions: Drug: Simvastatin 20 mg; Drug: Methotrexate 10 mg
- Methotrexate (Active Comparator): Methotrexate 10 mg once a week for 6 months
  Interventions: Drug: Methotrexate 10 mg

INTERVENTIONS:
Drug: Simvastatin 20 mg — improvement of disease activity
  Arms: Simvastatin & Methotrexate
Drug: Methotrexate 10 mg — improvement of disease activity

SUMMARY:
The objective of the study is to compare the efficacy of combination of Methotrexate and Statins with Methotrexate alone in the treatment of Rheumatoid Arthritis. It is hypothesized that adding statins to methotrexate for treatment of rheumatic arthritis will significantly suppress the disease activity as compared to methotrexate alone.

DETAILED DESCRIPTION:
After approval from Board of Studies and IRB of King Edward Medical University, all patients fulfilling inclusion and exclusion criteria from out patient department and wards of Mayo Hospital Lahore will be selected and randomized to group A or group B by lottery method (using coin flipping method) with one group receiving combination of methotrexate and simvastatin and other group receiving simvastatin only. All patients will be given adequate dose of analgesics for pain relief. Informed consent will be obtained from the patient. Demographic information like name, age and sex, will also be obtained. DAS 28 scoring will be done at the time of presentation and will be noted. Patients will be followed at 1 month, 3 month and at 6 month. At each follow up DAS 28(ESR) score will be calculated using DAS 28 calculator. All this information will be recorded on predesigned proforma (attached).

ELIGIBILITY:
Inclusion Criteria:

* All patients between ages 18 years and above
* Gender- Both male and female
* Fulfilling 2010 ACR/EULAR criteria of Rheumatoid arthritis with active inflammatory disease defined by DAS 28 score >2.6,
* Normal serum cholesterol level.

Exclusion Criteria:

* Already diagnosed patients of Diabetes mellitus.
* Use of steroids greater than 4 weeks of duration or intra articular steroid injection within 4 weeks of study.
* Statin therapy in last three months.
* Statin intolerant patient.
* Elevated Creatinine Phosphokinase more than twice the upper limit of normal range.
* Diagnosed case of Chronic liver disease or abnormal liver functions (transaminases > 2 times the upper limit of normal range) before the start of treatment or during follow-up.
* High serum Creatinine level
* Pregnancy and breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of drugs defined by improvement in Disease Activity Score 28 (DAS28) | 6 months
  In Rheumatoid arthritis, DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. A DAS 28 below the value of 2.6 is interpreted as Remission/improvement

SECONDARY OUTCOMES:
Adverse Drug Reaction | 6 months
  Adverse event reported against any of the intervention under study

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Rathore, FCPS, Principal Investigator — Associate Professor
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam SM, Kidwai AA, Jafri SR, Qureshi BM, Sami A, Qureshi HH, Mirza H. Epidemiology of rheumatoid arthritis in a tertiary care unit, Karachi, Pakistan. J Pak Med Assoc. 2011 Feb;61(2):123-6. PMID 21375157
- [Result] Wells G, Becker JC, Teng J, Dougados M, Schiff M, Smolen J, Aletaha D, van Riel PL. Validation of the 28-joint Disease Activity Score (DAS28) and European League Against Rheumatism response criteria based on C-reactive protein against disease progression in patients with rheumatoid arthritis, and comparison with the DAS28 based on erythrocyte sedimentation rate. Ann Rheum Dis. 2009 Jun;68(6):954-60. doi: 10.1136/ard.2007.084459. Epub 2008 May 19. PMID 18490431
- [Result] Mowla K, Rajai E, Ghorbani A, Dargahi-Malamir M, Bahadoram M, Mohammadi S. Effect of Atorvastatin on the Disease Activity and Severity of Rheumatoid Arthritis: Double-Blind Randomized Controlled Trial. J Clin Diagn Res. 2016 May;10(5):OC32-6. doi: 10.7860/JCDR/2016/16538.7814. Epub 2016 May 1. PMID 27437268
- [Result] Das S, Mohanty M, Padhan P. Outcome of rheumatoid arthritis following adjunct statin therapy. Indian J Pharmacol. 2015 Nov-Dec;47(6):605-9. doi: 10.4103/0253-7613.169585. PMID 26729950
- [Result] Aoki C, Nakano A, Tanaka S, Yanagi K, Ohta S, Jojima T, Kasai K, Takekawa H, Hirata K, Hattori Y. Fluvastatin upregulates endothelial nitric oxide synthase activity via enhancement of its phosphorylation and expression and via an increase in tetrahydrobiopterin in vascular endothelial cells. Int J Cardiol. 2012 Apr 5;156(1):55-61. doi: 10.1016/j.ijcard.2010.10.029. Epub 2010 Nov 18. PMID 21093076
- [Result] Abeles AM, Marjanovic N, Park J, Attur M, Chan ES, Al-Mussawir HE, Dave M, Fisher MC, Stuchin SA, Abramson SB, Pillinger MH. Protein isoprenylation regulates secretion of matrix metalloproteinase 1 from rheumatoid synovial fibroblasts: effects of statins and farnesyl and geranylgeranyl transferase inhibitors. Arthritis Rheum. 2007 Sep;56(9):2840-53. doi: 10.1002/art.22824. PMID 17763406
- [Result] Lazzerini PE, Lorenzini S, Selvi E, Capecchi PL, Chindamo D, Bisogno S, Ghittoni R, Natale MR, Caporali F, Giuntini S, Marcolongo R, Galeazzi M, Laghi-Pasini F. Simvastatin inhibits cytokine production and nuclear factor-kB activation in interleukin 1beta-stimulated synoviocytes from rheumatoid arthritis patients. Clin Exp Rheumatol. 2007 Sep-Oct;25(5):696-700. PMID 18078616
- [Result] Gazzerro P, Proto MC, Gangemi G, Malfitano AM, Ciaglia E, Pisanti S, Santoro A, Laezza C, Bifulco M. Pharmacological actions of statins: a critical appraisal in the management of cancer. Pharmacol Rev. 2012 Jan;64(1):102-46. doi: 10.1124/pr.111.004994. Epub 2011 Nov 21. PMID 22106090
- [Result] Agrawal S, Misra R, Aggarwal A. Autoantibodies in rheumatoid arthritis: association with severity of disease in established RA. Clin Rheumatol. 2007 Feb;26(2):201-4. doi: 10.1007/s10067-006-0275-5. Epub 2006 Mar 30. PMID 16572283
- [Result] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Result] Dowman B, Campbell RM, Zgaga L, Adeloye D, Chan KY. Estimating the burden of rheumatoid arthritis in Africa: A systematic analysis. J Glob Health. 2012 Dec;2(2):020406. doi: 10.7189/jogh.02.020406. PMID 23289081